CLINICAL TRIAL: NCT05106816
Title: The Effects of Vibrotactile Stimulation (Not Impossible Vibrohealth) on Motor Control and Symptoms in Patients With Movement Disorders
Brief Title: The Effects of Vibrotactile Stimulation in Patients With Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Parkinson's Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202002167
Record Dates: First submitted 2021-10-12; First posted 2021-11-04 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia
Keywords: Parkinson Disease; Essential tremor; Dystonia; Vibrotactile stimulation
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia

STUDY DESIGN:
Intervention Model Description: All participants will undergo tremor measurements and perform motor control tasks at baseline and during continuous vibratory stimulation and sham stimulation.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research subjects will be blinded regarding stimulation or sham and specific stimulation settings. Walking will be scored by a blinded rater for number of freezing episodes and walking completion time in seconds in the timed up and go task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vibrotactile Continuous stimulation (Experimental): Continuous stimulation
  Interventions: Other: skin surface vibration
- Vibrotactile Intermittent stimulation (Experimental): Intermittent stimulation
  Interventions: Other: skin surface vibration
- Vibrotactile Sham (Sham Comparator): Sham stimulation
  Interventions: Other: light skin surface vibration- SHAM

INTERVENTIONS:
Other: skin surface vibration — This study will use four vibrating devices worn on each of the limbs. The devices are paired with a cell phone application (to be used solely by research investigators) that adjusts the vibration settings. The intensity of the vibration produced by the device is far less than that produced by commercially available massagers used for relaxation using similar technology. The sensor in the device is a tri-axial accelerometer and gyroscope that measures position using the same technology as smartphones.
  Arms: Vibrotactile Continuous stimulation; Vibrotactile Intermittent stimulation
Other: light skin surface vibration- SHAM — This study will use four vibrating devices worn on each of the limbs. The devices are paired with a cell phone application (to be used solely by research investigators) that adjusts the vibration settings. The intensity of the vibration produced by the device is far less than that produced by commercially available massagers used for relaxation using similar technology. The sensor in the device is a tri-axial accelerometer and gyroscope that measures position using the same technology as smartphones. Worn at the lowest frequency will simulate the active arms with no potential change in symptoms.
  Arms: Vibrotactile Sham

SUMMARY:
Vibration applied to the skin has been anecdotally reported to potentially improve motor control in patients with movement disorders including Parkinson's disease, however few devices have been studied formally. In this study, the investigators will test the effect of skin surface vibration applied non-invasively to patients with movement disorders to determine if there are any beneficial effects on common tasks of motor control and/or abnormal motor symptoms in patients with Parkinson's disease (PD), essential tremor (ET), and dystonia.

DETAILED DESCRIPTION:
This study is to evaluate the feasibility, reliability, and clinical effects of Non-invasive vibrotactile stimulation (VTS) on basic tasks of motor control and on the motor symptoms of patients with movement disorders. VTS Settings will include continuous stimulation, intermittent stimulation during walking, and sham stimulation.

The investigators will recruit 30 patients with PD who are between the ages of 18-80 years old and independently living in the community. The investigators will additionally recruit up to 5 patients with ET and up to 5 patients with dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 and able to provide informed consent.
* Have a diagnosis of Parkinson's disease, essential tremor, or cervical dystonia made by a movement disorders specialist.
* Medically optimized without planned medication changes for the duration of the study.
* For patients with ET, they will have a score of at least 2 on items 5 and 6 of the Fahn-Tolosa-Marin (FTM) Tremor Rating Scale.
* For patients with dystonia, they will have abnormal dystonic postures of the head and not isolated head tremor

Exclusion Criteria:

* The presence of additional neurologic diseases, that might confound testing or the coexistence of PD and ET together (action tremor that was present prior to the development of parkinsonism).
* Symptoms of peripheral neuropathy at the wrist (reduced vibratory, pinprick, or temperature sensation)
* Montreal cognitive assessment (MoCA) score < 20 or previously documented dementia
* Unable to walk without a walking aid (e.g. cane, stick, walker)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Quantitative Tremor Assessment | Baseline up to immediately after the sham intervention
  An external accelerometer will be adhered to the skin of the dorsum of the hand and will be used to quantify displacement of the hand due to tremor in the following conditions:
  * 1. Sitting at rest
  * 2. Sitting with both arms outstretched
  * 3. Sitting at rest while performing a distracting cognitive task
  * 4. Transition from rest to posture (arms held directly in front of patient) for 10 seconds

SECONDARY OUTCOMES:
Functional Dexterity Task (FDT) | Baseline up to immediately after the sham intervention
  Functional Dexterity Task (FDT): The FDT is a pegboard assessment of manual dexterity.
Reaction time task | Baseline up to immediately after the sham intervention
  Subjects will look at a central fixation symbol on computer screen and press a computer keyboard/mouse button when the GO signal appears. The time between the onset of the fixation cross and the green GO signal will vary so that the onset of the GO signal will not be predictable. The time between appearance of the GO signal and recorded keyboard response will be recorded as reaction time
Timed-up-and-go (TUG) gait task | Baseline up to immediately after the sham intervention
  Subjects are asked to stand up from a chair, walk 3 meters to a horizontal line marked with red tape on the floor, turn around, walk back and sit down, at a comfortable pace. this task will be performed on an the instrumented mat that measures gait characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Hess, MD, Principal Investigator — Norman Fixel Institute for Neurological Diseases, University of Florida
Locations (1):
- Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data will be published, but no PHI will be made available.

REFERENCES:
- [Background] Charcot JM. Vibratory therapeutics.--The application of rapid and continuous vibrations to the treatment of certain diseases of the nervous system. 1892. J Nerv Ment Dis. 2011 Nov;199(11):821-7. doi: 10.1097/NMD.0b013e31823899bc. No abstract available. PMID 22048131
- [Background] Gassner H, Janzen A, Schwirtz A, Jansen P. Random Whole Body Vibration over 5 Weeks Leads to Effects Similar to Placebo: A Controlled Study in Parkinson's Disease. Parkinsons Dis. 2014;2014:386495. doi: 10.1155/2014/386495. Epub 2014 Oct 13. PMID 25371843
- [Background] Haas CT, Turbanski S, Kessler K, Schmidtbleicher D. The effects of random whole-body-vibration on motor symptoms in Parkinson's disease. NeuroRehabilitation. 2006;21(1):29-36. PMID 16720935
- [Background] Jobges EM, Elek J, Rollnik JD, Dengler R, Wolf W. Vibratory proprioceptive stimulation affects Parkinsonian tremor. Parkinsonism Relat Disord. 2002 Jan;8(3):171-6. doi: 10.1016/s1353-8020(01)00016-5. PMID 12039427
- [Background] Kapur SS, Stebbins GT, Goetz CG. Vibration therapy for Parkinson's disease: Charcot's studies revisited. J Parkinsons Dis. 2012;2(1):23-7. doi: 10.3233/JPD-2012-12079. PMID 23939405

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT05106816/Prot_SAP_000.pdf